CLINICAL TRIAL: NCT06312540
Title: Longitudinal Study of Biomarkers for Personalized Post-Stroke Rehabilitation
Brief Title: PERSonalized rObotic NeurorehAbilitation for Stroke Survivors
Acronym: PERSONA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Principal Investigator, Carmelo Chisari, Head of Neurorehabilitation Unit, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: PERSONA; 15397/2018 (Other Grant/Funding Number: Tuscany Region - Bando FAS)
Record Dates: First submitted 2024-02-19; First posted 2024-03-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Stroke Acute
Keywords: Stroke recovery; Biomarkers; EEG; Machine Learning; Upper extremities
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim is to carry out a first clinical study, to expand existing knowledge about the neurophysiological mechanisms underlying post-stroke recovery. The information acquired during this phase will be used as building blocks to develop customized protocols. Understanding the mechanisms underlying stroke-induced motor deficits and motor recovery is mandatory to improve clinicians; ability to guide the repair of the affected neural structures. The motor system comprises a network of cortical and subcortical areas interacting via excitatory and inhibitory circuits, thereby governing motor behaviour. Stroke lesions cause neural dysfunction both at the lesion site and in remote brain regions. Abnormal interactions among cortical regions within the motor network contribute to the motor impairment after stroke. Longitudinal analysis of neural activity and connectivity can help to understand the pathophysiology mechanisms underlying functional impairment and recovery after stroke. Analysis of the data will try to extract biomarkers of plasticity and recovery that will be used to design customized therapeutic interventions.

DETAILED DESCRIPTION:
Consecutive stroke patients admitted to the Stroke Unit will be enrolled. Both ischaemic and hemorrhagic strokes above 18-years of age will be recruited. A dedicated encrypted database will be developed, and the following items will be collected: age, sex, aetiology of stroke, TOAST classification, Modified Rankin Scale before stroke and at the discharge from the Stroke Unit and after 3 months from the stroke (in survivors), NIHSS at the onset, at the discharge from the Stroke Unit, and after 3 months from the stroke (in survivors), neuroimaging studies at the onset (CT, AngioCT, MRI) and the follow up, acute treatment (for ischaemic strokes, fibrinolysis, primary or rescue thrombectomy, standard care), comorbidity (diabetes, hypertension, smoking habits, heart disease, atrial fibrillation, etc), biochemical and genetic biomarkers from blood and urine. The clinical and biochemical section of our database will include "yes or no" dichotomic items agreed by all groups in a preliminary consensus phase, specifically designed to define the clinical features known to be relevant in strokes.

ELIGIBILITY:
Inclusion Criteria:

* unilateral motor deficit (with or without other stroke- related symptoms or signs)
* radiological evidence of unilateral, supratentorial cerebral ischemic lesion (or lesions) in the same arterial territory
* stroke occurred in the last 4 days
* absent or slight disability before stroke estimated by a modified Rankin Scale 0-2

Exclusion Criteria:

* history of severe cognitive impairment
* psychiatric comorbidities
* end-stage organic diseases like cardiopulmonary, hepatic, renal failure, neoplasms, and whatever condition that could strongly reduce life expectation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke survivors
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Brain activity | 36 months
  Electroencephalography (EEG) power spectrum analysis
Functional evaluation | 36 months
  Fugl-Meyer Upper Limb (0-66)

SECONDARY OUTCOMES:
Clinical scale | 36 months
  Motricity Index (0-100)
  Wolf Motor Function Test
Spasticity assessment | 36 months
  Modified Ashworth Scale (0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Chisari, Medical, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- AOUPisana, Pisa, Pi, Italy

IPD SHARING:
Plan to Share IPD: No